CLINICAL TRIAL: NCT06613061
Title: Breathing Exercise Women Receiving Brachytherapy
Brief Title: Effects of Breathing Exercises on Pain, Fatigue, and Anxiety Levels in Women Receiving Brachytherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Neşe Uysal, Director, Amasya University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-NU-689
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Exercise
Keywords: radiothreapy
MeSH Terms: conditions — Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (breathing exercise) (Experimental): The researcher has a breathing exercise certificate. In our study, the breathing exercise application consists of three stages: box breathing, sigh breathing and diaphragm breathing.
  Patients will be asked to continue the breathing exercise application for 2 weeks and will be reminded to do the breathing exercises. Box and sigh breathing will be done 3 times a day (morning, noon and evening) every day for 2 weeks. Diaphragm breathing exercise will be applied for 2 minutes in the first week and 4 minutes in the second week.
  Interventions: Other: Breathing exercise
- Control (No Intervention): The control group will receive standard care. No intervention will be applied to these patients during the follow-up period, only data collection forms will be applied. Data collection forms will be collected in the same time period as the intervention group.

INTERVENTIONS:
Other: Breathing exercise — The researcher has a breathing exercise certificate. In our study, the breathing exercise application consists of three stages: box breathing, sigh breathing and diaphragm breathing.
  Patients will be asked to continue the breathing exercise application for 2 weeks and will be reminded to do the breathing exercises. Box and sigh breathing will be done 3 times a day (morning, noon and evening) every day for 2 weeks. Diaphragm breathing exercise will be applied for 2 minutes in the first week and 4 minutes in the second week.
  Arms: Experimental (breathing exercise)

SUMMARY:
Breathing exercises are one of the most useful techniques to reduce stress and anxiety. The aim of this study is to determine the effects of breathing exercises on pain, anxiety and fatigue in patients receiving brachytherapy treatment.

DETAILED DESCRIPTION:
Introduction: Breathing exercises are one of the most useful techniques to reduce stress and anxiety.

Objective: The aim of this study is to determine the effects of breathing exercises on pain, anxiety and fatigue in patients receiving brachytherapy treatment.

Method: The sample of the study will consist of 56 women who applied to the Brachytherapy Unit of a training and research hospital. The research data will be collected using the Introductory Information Form, Numerical Pain Scale, Beck Anxiety Inventory and Piper Fatigue Scale. Although studies have been conducted in different areas regarding breathing exercises, no study has been found in our country regarding the effects of breathing exercises on patients receiving brachytherapy. Therefore, this study will determine the effects of breathing exercises on pain, anxiety and fatigue in patients receiving brachytherapy treatment and contribute to the literature.

Conclusion: It is thought that breathing exercises will be beneficial in reducing physical and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being willing to participate in the study
* Being able to speak and understand Turkish

Exclusion Criteria:

* Having a malignancy related to the respiratory system (bronchus or lung)
* Having chest pain
* Having done box breathing and diaphragm breathing exercises/receiving training before
* Having cognitive dysfunction
* Not giving consent to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Numerical pain scale | Two week
  Numerical pain scale: The numerical pain scale is a one-dimensional scale and the expressions "no pain" and "unbearable pain" are located at both ends of the figure. There are values between 0-10 on the scale at equal intervals and the patient marks them according to the level of pain.The scale scores between 0-10. The high total score indicates the high pain level experienced by the person.
Beck Anxiety Inventory | Two week
  The Beck Anxiety Inventory (BAI) is a Likert-type assessment scale consisting of 21 items and scored between 0-3, designed to measure the frequency of anxiety symptoms experienced by the individual. Individuals rate each item by giving a score between 0-3 to determine how uncomfortable they have felt "over the past week, including the day of the application". The scale scores between 0-63. The high total score indicates the high level of anxiety experienced by the person
Piper Fatigue Scale | Two week
  Piper Fatigue Scale (PFS): The PFS consists of 22 questions and evaluates fatigue perception subjectively. It has four sub-dimensions: the behavior/severity sub-dimension, which evaluates the effect and severity of fatigue on daily life activities; the affective sub-dimension, which covers the emotional meaning attributed to fatigue; the sensory sub-dimension, which reflects the mental, physical and emotional symptoms of fatigue; and the cognitive/spiritual sub-dimension, which reflects the degree to which fatigue affects cognitive functions and mood. The total score of the scale varies between 0 and 10. A score of 0 indicates no fatigue, 1-3 indicates mild fatigue, 4-6 indicates moderate fatigue, and 7-10 indicates severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)